CLINICAL TRIAL: NCT05355532
Title: Identification of Genetic Determinants of the Coronary Microvascular Obstruction Development in Percutaneous Coronary Interventions
Brief Title: Genetic Determinants of the Coronary Microvascular Obstruction in PCI
Status: Completed | Type: Observational
Sponsor: Privolzhsky Research Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: CMVO-SNP-2022
Record Dates: First submitted 2022-04-24; First posted 2022-05-02 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-05

CONDITIONS: Myocardial Infarction; No-Reflow Phenomenon
Keywords: coronary microvascular obstruction; no-reflow phenomenon; myocardial infarction; percutaneous coronary intervention; single nucleotide polymorphism; genetics
MeSH Terms: conditions — Myocardial Infarction; No-Reflow Phenomenon

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- "CMVO+" (patients has presented CMVO in PCI): Patients with 1 type MI that has presented CMVO in emergency PCI.
  Interventions: Genetic: different variants of SNPs that may be associated with the coronary microvascular obstruction development
- "CMVO-" (patients hasn't presented CMVO in PCI): Patients with 1 type MI that hasn't presented CMVO in emergency PCI.
  Interventions: Genetic: different variants of SNPs that may be associated with the coronary microvascular obstruction development

INTERVENTIONS:
Genetic: different variants of SNPs that may be associated with the coronary microvascular obstruction development — Some variants of SNPs determine endothelial function, microcirculation, hemostasis, and inflammation in MI patients. They may be associated with the development of coronary microvascular obstruction during emergency PCI. A link between the different SNPs and the CMVO development will be established. SNP will be determined by real-time polymerase chain reaction with high-resolution melting curve analysis using TaqMan fluorescent probes.

SUMMARY:
Myocardial infarction (MI) remains one of the most common causes of death. Percutaneous coronary intervention (PCI) is the main treatment option to restore blood flow through the infarction-related coronary artery (IRA) in MI patients. Performing PCI significantly reduces mortality, but in 5-10% cases, PCI is complicated by the development of coronary microvascular obstruction (CMVO, "no-reflow"). CMVO is defined as the absence of adequate myocardial perfusion, despite the restoration of the IRA lumen. The development of CMVO significantly worsens the prognosis and increases mortality.

CMVO has a complex pathogenesis and is development due to following mechanisms: distal microembolism, ischemia-reperfusion injury, persistent endothelial dysfunction, and individual predisposition. These mechanisms can be implemented simultaneously and have different severity. The most significant predictors of CMVO occurrence are: age, time from pain onset to reperfusion, severity of acute heart failure, ineffective thrombolytic therapy, collateral blood flow according to the Rentrop classification, severity of IRA thrombosis according to Thrombolysis in Myocardial Infarction (TIMI) thrombus grade, initial IRA blood flow according to TIMI flow grade, implantation of 3 or more stents, direct IRA stenting, neutrophil and blood glucose levels.

Difficulties in CMVO predicting are caused by the pathogenetic heterogeneity of this complication. Even the best models are moderately accurate. This can be explained by the fact that the models don't use genetic factors that determine endothelial function, microcirculation, hemostasis, and inflammation. Identification of the genetic determinants of the CMVO development can help create a new diagnostic system for CMVO predicting.

DETAILED DESCRIPTION:
The aim of the study to identify the genetic determinants of the coronary microvascular obstruction development during percutaneous coronary interventions in myocardial infarction patients. The study investigates the role of some variants of single nucleotide polymorphism (SNP) as predictors of CMVO development. Selected SNPs that are associated with the mechanisms of CMVO development (according to literature). Hypothesis: selected SNPs are independent genetic predictors of the development of CMVO during PCI in MI patients.

Study design: matched case-control study. Sample size: 80 patients. Patients must have inclusion criteria, haven't exclusion criteria, and sign an informed consent. Division into 2 groups in the ratio 1:1. Group 1 (CMVO+): 40 patients with MI who were detected the CMVO after PCI. The second group (CMVO-, control): 40 patients with MI who weren't detected CMVO after PCI. Groups are matched by sex and age. The sample size (80 patients) was determined in accordance with the following parameters: alpha error - 5%, study power - 80%, group size ratio - 1:1, minimum odds ratio for detection - 4.0, prevalence SNP in the population - 12-69% (average 50%).

CMVO (no-reflow) is defined as inadequate myocardial perfusion after successful mechanical restoration of blood flow through the IRA (according to the 2017 European Society of Cardiology STEMI guidelines). CMVO criteria (there must be at least one criterion): 1) IRA blood flow is less than 3 points according to TIMI flow grade; 2) myocardial perfusion less than 2 points according to Myocardial blush grade (MBG). Other causes of IRA obstruction (spasm, dissection, thromboembolism) must be excluded.

Research stages: 1) assessment of inclusion / exclusion criteria; 2) signing informed consent; 3) taking blood for genetic analysis (performed in the operating room immediately after PCI); 4) processing of blood samples and their transportation to the laboratory; 5) filling out the patient's register card (contains information about the treatment and outcomes); 6) performing genetic analysis; 7) statistical processing of the obtained results.

The registration card is filled in at the end of hospitalization. Purpose: 1) comparison of SNP variants and outcomes; 2) multivariate analysis of SNP variants and other CMVO predictors. The card contains the following data: information about PCI, risk factors for the CMVO development, laboratory data (general blood count, biochemical blood test, etc.), examination data (ECG, ECG monitoring, echocardiography, six-minute walk test), information about complications and outcomes. These laboratory tests and instrumental studies are used in accordance with routine hospital protocols for the treatment of MI patients (the using is not associated with the investigation).

Venous peripheral blood is used for genetic testing. Blood sampling is performed directly in the operating room after PCI. Selected SNPs from the "CardioGenetics Hypertension" panel, "CardioGenetics Thrombophilia" panel and "Genetics of Folate Metabolism" panel from the "DNA-Technology" company (Russia). Also used a set of reagents for the detection of Lys198Asn polymorphism in the EDN1 gene "SNP-Express-Cardiogenetics RT" from "Litekh" Company (Russia). SNPs are determined by real-time polymerase chain reaction with high resolution melt curve analysis using TaqMan fluorescent probes. The following SNPs are analyzed (SNP identifier and gene): rs4961 (ADD1); rs699 и rs4762 (AGT); rs5186 (AGTR1); rs1403543 (AGTR2); rs1799998 (CYP11B2); rs5443 (GNB3); rs2070744 и rs1799983 (eNOS); rs1799963 (F2); rs6025 (F5); rs6046 (F7); rs5985 (F13); rs1800790 (FGB); rs1126643 (ITGA2-α2); rs5918 (ITGB3-β3); rs1799762 (PAI-1); rs1801133 (MTHFR); rs1801131 (MTHFR); rs1805087 (MTR); rs1801394 (MTRR); rs5370 (EDN1).

Expected results: it will be proved or disproved that some variants of SNP are independent predictors of the development of CMVO during PCI in patients with myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

1. informed consent to participate in the study;
2. male or female 18 years of age or older;
3. type 1 ST-segment elevation MI (according to the criteria of the fourth universal definition of myocardial infarction and current clinical guidelines);
4. blood sampling in the operating room (immediately after PCI) and signing the informed consent;
5. for the "CMVO+" group: CMVO because of PCI (CMVO is registered according to the criteria from the European Society of Cardiology clinical guidelines);
6. for the "CMVO-" group: absence of CMVO after PCI; patient should compliance by sex and age (±5 years) with pair in the "CMVO+" group.

Exclusion Criteria:

1. late admission (more than 48 hours from the onset of anginal pain) or early post-infarction angina pectoris;
2. not 1 type MI;
3. complications during PCI (dissection, perforation or acute intraoperative thrombosis of the IRA);
4. death during PCI, not due to the CMVO development;
5. concomitant terminal pathology (not associated with MI) with a life expectancy less than 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with 1 type MI after emergency PCI
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Pochinka, MD, Study Chair — Privolzhsky Research Medical University
Locations (2):
- Russia (2):
  - City Clinical Hospital No. 13 of the Avtozavodsky District of Nizhny Novgorod, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Central Research Laboratory of the Privolzhsky Research Medical University, Nizhny Novgorod, Nizhny Novgorod Oblast

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frolov AA, Pochinka IG, Shakhov BE, Mukhin AS, Frolov IA, Barinova MK, Sharabrin EG. Using an Artificial Neural Network to Predict Coronary Microvascular Obstruction (No-Reflow Phenomenon) during Percutaneous Coronary Interventions in Patients with Myocardial Infarction. Sovrem Tekhnologii Med. 2021;13(6):6-13. doi: 10.17691/stm2021.13.6.01. Epub 2021 Dec 28. PMID 35265354
- [Result] Frolov A.A., Pochinka I.G., Kuzmichev K.V., Shchelchkova N.A., Pershin V.I., Maksimova N.S., Budkina M.L., Predeina I.V., Mukhin A.S. Genetic markers of endothelial dysfunction as predictors of coronary microvascular obstruction in endovascular treatment of myocardial infarction. Cardiology: News, Opinions, Training. 2025; 13 (1): 22-30. DOI: 10.33029/2309-1908-2025-13-1-22-30
- [Result] Pochinka IG, Shchelchkova NA, Frolov AA, Pershin VI, Maksimova NS, Kuzmichev RV, Budkina ML, Predeina IV, inventors. Privolzhsky Research Medical University, assignee. Method of diagnosing genetic predisposition to development of phenomenon of coronary microvascular obstruction during percutaneous coronary interventions in patients with myocardial infarction with ST segment elevation. Russian Federation patent RU 2,811,933. 2023 Oct 26.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | "CMVO+" (Patients Has Presented CMVO in PCI) | "CMVO-" (Patients Hasn't Presented CMVO in PCI)
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | "CMVO+" (Patients Has Presented CMVO in PCI) | "CMVO-" (Patients Hasn't Presented CMVO in PCI) | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [60 to 73] | 65 [61 to 71] | 65 [60 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 29 | 29 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 40 | 80
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Hospital Mortality Rate
Description: Death during index hospitalization.
Time Frame: up to 7-15 days after PCI
Measure: Count of Participants; unit: Participants
Arm/Group | "CMVO+" (Patients Has Presented CMVO in PCI) | "CMVO-" (Patients Hasn't Presented CMVO in PCI)
Number analyzed (Participants) | 40 | 40
Participants | 6 | 2

2. Secondary Outcome: Left Ventricle Ejection Fraction
Description: Echo-cardiography, four-chamber projection, Simpson's method.
Time Frame: 7-10 day after PCI
Measure: Median (Inter-Quartile Range); unit: ejection fraction percent
Arm/Group | "CMVO+" (Patients Has Presented CMVO in PCI) | "CMVO-" (Patients Hasn't Presented CMVO in PCI)
Number analyzed (Participants) | 40 | 40
ejection fraction percent | 47 [38 to 51] | 50 [43 to 53]

3. Secondary Outcome: Six-minute Walk Test
Description: Distance in meters that a patient can walk in 6 minutes. Based on the test, the class of chronic heart failure according to New York Heart Association (NYHA) classification is determined.
Time Frame: 7-10 day after PCI
Measure: Median (Inter-Quartile Range); unit: meters in 6 minutes
Arm/Group | "CMVO+" (Patients Has Presented CMVO in PCI) | "CMVO-" (Patients Hasn't Presented CMVO in PCI)
Number analyzed (Participants) | 40 | 40
meters in 6 minutes | 395 [320 to 443] | 425 [380 to 465]

4. Secondary Outcome: N-terminal Pro-brain Natriuretic Peptide
Description: Level of N-terminal pro-brain natriuretic peptide in pg/ml
Time Frame: 7-10 day after PCI
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | "CMVO+" (Patients Has Presented CMVO in PCI) | "CMVO-" (Patients Hasn't Presented CMVO in PCI)
Number analyzed (Participants) | 40 | 40
pg/ml | 1171 [506 to 2071] | 530 [333 to 916]

5. Secondary Outcome: Ventricular Fibrillation
Description: Ventricular fibrillation during index hospitalization
Time Frame: up to 7-15 days after PCI
Measure: Count of Participants; unit: Participants
Arm/Group | "CMVO+" (Patients Has Presented CMVO in PCI) | "CMVO-" (Patients Hasn't Presented CMVO in PCI)
Number analyzed (Participants) | 40 | 40
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 7-15 days after PCI
Description: a standard definition of adverse events was used
Arm/Group | "CMVO+" (Patients Has Presented CMVO in PCI) | "CMVO-" (Patients Hasn't Presented CMVO in PCI)
All-Cause Mortality (participants affected / at risk) | 6/40 | 2/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT05355532/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT05355532/SAP_001.pdf
  • Informed Consent Form (2022-04-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT05355532/ICF_002.pdf